CLINICAL TRIAL: NCT05086939
Title: Phase III, Multicenter, Randomized, Open-label Clinical Trial Comparing Treatment with Allogeneic Mesenchymal Cells Versus Autologous Mesenchymal Cells and Versus Active Control with Hyaluronic Acid in Patients with Knee Osteoarthritis
Brief Title: Multicenter Clinical Trial Comparing Treatment with Allogeneic Mesenchymal Cells Versus Autologous Mesenchymal Cells and Versus Active Control with Hyaluronic Acid in Patients with Knee Osteoarthritis.
Acronym: ARTROCELL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Spanish Clinical Research Network - SCReN (Network); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTROCELL; 2019-002446-21 (EudraCT Number); 2024-514545-11-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-05; First posted 2021-10-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, Open-label, Clinical Trial comparing 3 active treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Autologous Mesenchymal Stromal Cells (MSC) (Experimental): Treatment with 40 millions of autologous autologous adult mesenchymal stem cells from expanded bone marrow administered intra-articularly.
  Interventions: Drug: Autologous MSCs
- Allogenic Mesenchymal Stromal Cells (MSC) (Experimental): Treatment with 40 millions of adult allogeneic expanded bone marrow mesenchymal stem cells administered intra-articularly.
  Interventions: Drug: Allogenic MSCs
- Active Control (Active Comparator): Hyaluronic Acid 60mg/3ml administered intra-articularly.
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: Autologous MSCs — Intra-articular injection 40 million/4 ml.
  Arms: Autologous Mesenchymal Stromal Cells (MSC)
Drug: Allogenic MSCs — Intra-articular injection 40 million/4 ml.
  Arms: Allogenic Mesenchymal Stromal Cells (MSC)
Drug: Hyaluronic Acid — Intra-articular injection 60mg / 3 ml .
  Other Names: Hyaluronic Acid 20 mg/ml
  Arms: Active Control

SUMMARY:
Phase III, multicenter, randomized, open-label, multicenter clinical trial comparing treatment with allogeneic mesenchymal cells versus autologous mesenchymal cells and versus active control with hyaluronic acid in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Gonarthrosis grade 2, 3 or 4 of Kellgren and Lawrence (Kellgren & Lawrence, 1957) assessed by two observers.
2. Chronic painful knee of mechanical characteristics.
3. Absence of local or systemic septic process.
4. Hemat imetric and biochemical analysis without significant alterations that contraindicate the treatment.
5. Written informed consent of the patient.
6. The patient is able to understand the nature of the study.
7. Body Mass Index 20-35 Kg/m2.

Exclusion Criteria:

1. Patient < 18 years old, or legally dependent.
2. Patient > 75 years old.
3. Congenital or developmental diseases that translate malformation and / or significant deformations of the knee (varus>10º; valgus>20º) and condition difficulties of application and evaluation of the results.
4. Pregnant or breastfeeding women.
5. Neoplastic disease.
6. Intra-articular infiltration of any drug in the 3 months prior to study inclusion.
7. Concurrent participation in another clinical trial or treatment with another investigational product within 30 days prior to study enrollment.
8. Allergy to gentamicin (antibiotic used in the cell culture process ).
9. Other diseases or circumstances that compromise participation in the study according to medical criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Range of motion. | 12 months
  Evaluation of clinical-functional response using Joint range-of-motion evaluation (Flexion score 0º-140º / Extension score -140º-0º / Hyperextension: positive degrees from 0).
Pain self-assessment. | 12 months
  Evaluation of pain using Visual Analogue Scale (VAS) (Pain self-assessment score range from 0 -no pain- to 10 -maximum-).
Knee Osteoarthritis. | 12 months
  Evaluation of Knee Osteoarthritis using Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) [measures five items for pain (score range from 0 -no pain- to 20 -maximum-), two for stiffness (score range from 0-no stiffness- to 8 -maximum-), and 17 for functional limitation (score range from 0 -no limitation- to 68 -maximum-)]
Functional response. | 12 months
  Evaluation of functional response using Lequesne Algofunctional Index (score range from 0 to 24). It includes measures of pain (5 questions), walking distance (1 question) and activities of daily living (4 questions) with separate versions for the hip and knee. The scores for each question are summed to obtain a combined score of disease severity. Scores 1 to 4 are classified as mild osteoarthrosis; 5 to 7, moderate; 8 to 10, severe; 11 to 13, very severe; and 14 and above, extremely severe.
X-ray changes of osteoarthritis. | 12 months
  Radiological response using Kellgren and Lawrence classification system (grade from 0 to 4):
  * grade 0 (none): definite absence of x-ray changes of osteoarthritis.
  * grade 1 (doubtful): doubtful joint space narrowing and possible osteophytic lipping.
  * grade 2 (minimal): definite osteophytes and possible joint space narrowing.
  * grade 3 (moderate): moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends.
  * grade 4 (severe): large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends.
Radiological response using nuclear magnetic resonance imaging. | 12 months
  Evaluation of radiological response using T2 mapping nuclear magnetic resonance imaging (screening visit global mean of T2 values versus 12 months visit global mean of T2 values).

SECONDARY OUTCOMES:
Perceived general well-being. | 6, 12 and 24 months
  Evaluation of quality of life using Short Form-12 Health Survey questionnaire (SF12) [score range from 0 (the worst health status for that dimension) to 100 (the best health status)]
Feasibility assessment of a multicentre strategy production of both cell types with several Cell Production Units | 24 months
  Rate of products not conforming to the validation criteria in each arm of experimental treatment.
Evaluation of presence of adverse events related with investigational medical product (IMP). | 24 months
  Rate of adverse events and other pharmacovigilance parameters in the three treatment arms.
Evaluation of products obtained by genomic study and potency studies of the final products of all cell types (exploratory objective) | 30 days
  Studies of the cell product. In this exploratory objective, genomic studies will be carried out using RNA-seq and open array on the advanced therapy drugs manufactured in the study (both autologous and allogeneic), and a correlation will be made with clinical and biological parameters and with the response.
Evaluate induced changes in circulating cells of the immune system after cell treatment (exploratory objetive) | 30 days
  Evaluation of cell populations (NK cells, B cells, regulatory T cells, myeloid suppressor cells, T cell populations) by flow cytometry, prior to administration of cell therapy, at 7 days and 30 days.
  Evaluation of activation and inhibition markers in T lymphocytes (CD69, HLADR, CD137, PD1, LAG3 and TIM3) prior to administration of cell therapy, at 7 days and 30 days Population of inflammatory cytokines circulating in peripheral blood (Plex deB iorad -reference M50DKFADY), prior to administration of treatment, at 7 days and 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Sánchez-Guijo, Principal Investigator — IBSAL - University Hospital of Salamanca
Locations (8):
- Spain (8):
  - Hospital Clinic, Barcelona
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Clínica Universidad de Navarra, Pamplona
  - Complejo Asistencial Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No